CLINICAL TRIAL: NCT02142088
Title: A Clinical Study to Evaluate the Safety of the GlySure Continuous Intra-vascular Glucose Monitoring System, and Its Performance in Comparison to Intermittent Blood Glucose Monitoring in Adult Intensive Care Unit Patients
Brief Title: Comparative Study of GlySure Continuous Intra-vascular Glucose Monitoring and Intermittent Monitoring in Medical ICU
Acronym: MICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: GlySure (Industry)
Collaborators: Kentron (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014.01.CE
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Blood Glucose Monitoring in Medical ICU
Keywords: Glycaemic Control; Glucose Monitoring; Intravascular Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Glucose Monitoring (Other): Each patient will undergo simultaneous Glucose monitoring with 2 devices. One is GlySure's intervascular continuous measurement sensor (test device) introduced through a CVC, and the other measures glucose intermittently from repeated venous blood samples drawn through an indwelling ventflon style catheter
  Interventions: Device: GlySure Intravascular Continuous glucose monitoring sensor

INTERVENTIONS:
Device: GlySure Intravascular Continuous glucose monitoring sensor — Comparator device is an iSTAT device from Abbott Diagnostics
  Other Names: Devices not yet issued for study, so serial numbers not yet linked to study.

SUMMARY:
It has been shown that close control of blood glucose levels in the intensive care unit patient has benefits for patient morbidity and mortality rates as well as an impact upon discharge times. GlySure has previously completed an evaluation of its intra-vascular glucose monitoring system in patients in a surgical ICU environment after cardiac surgery. This study seeks to evaluate the same equipment being used in a wider range of patients with a range of underlying conditions who require treatment in medical ICU's. The GlySure device consists of a sensor that is placed into the patient's blood through a central venous catheter. It measures blood glucose levels continuously which allows for more rapid control of blood glucose levels to be achieved as compared to existing methods where blood samples are taken repeatedly every 15 minutes or so.

The study is designed to show that the sensor can be used for a protracted period of time, giving accurate results when compared to a reference technique using the i-STAT device. The investigators intend to show that the device performs safely for the required time within the ICU.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legal representative MUST be willing to sign an informed consent document
2. Patient is male or female aged 18 years or above
3. Patient requires a CVC to be inserted as part of disease management and treatment
4. Patient is expected to remain in the intensive care unit for at least 36 hours post enrolment to the study

Exclusion Criteria:

1. Patient or legal representative is unable to provide written informed consent
2. Patient who is pregnant
3. Patient who is currently being administered Mannitol and/or may require the administration of Mannitol whilst in the ICU
4. Patient with history of pulmonary embolism (PE)
5. Patient with history of thrombosis
6. Patient with known hyper-coagulation
7. Patient with known history of heparin hypersensitivity
8. Patient with history of heparin induced thrombocytopenia
9. Participation in a clinical study involving an unlicensed pharmaceutical product or device within the 3 months prior to enrolment in this study
10. Patient with known hypersensitivity/allergy to adhesive I.V. dressings such as 3M Tegaderm film or StatLock® devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Safety in Use | During ICU Stay, normally less than 7 days
  No Serious Adverse Events causally related to the device
MARD Score | During ICU stay, normally less than 7 days
  Average aggregate MARD to be below 10%, 95% of subjects to have a MARD of less than 25%